CLINICAL TRIAL: NCT02176811
Title: The Cross Sectional Study to Investigate the Plasma Betatrophin Levels in Non-alcoholic Fatty Liver Disease and Healthy Controls
Brief Title: Plasma Betatrophin Levels in Non-alcoholic Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Alper Sonmez, Associate Professor, Gulhane School of Medicine
Other Study IDs: GSM-052014
Record Dates: First submitted 2014-06-22; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Non-alcoholic Fatty Liver Disease; Betatrophin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-alcoholic Fatty Liver Disese: no treatment
- healthy controls: no treatment

SUMMARY:
The study searched for answers to two questions:

1-What are the plasma betatrophin levels in subjects with non-alcoholic fatty liver disease and healthy controls.

2. Is there any relationship between plasma betatropin levels and different stage of non-alcoholic fatty liver disease 2.Is there any relationship between plasma betatropin levels and metabolic parameters in subjects with non-alcoholic fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven non-alcoholic fatty liver disease

Exclusion Criteria:

* Taking any drugs
* >20 gr/day alcohol consumption
* chronic metabolic diseases
* morbid obesity

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Outpatient clinics of gastroenterology
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-06; Primary Completion 2013-06 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Plasma betatrophin levels in subjects with non-alcoholic fatty liver disease and healthy controls. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine Department of Endocrinology and Metabolism, Ankara, Turkey (Türkiye)